CLINICAL TRIAL: NCT01622920
Title: Preliminary Clinical Study of Ultrasound to Measure Enamel Thickness
Acronym: UMET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Khalid Sindi, Mr, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UMET
Record Dates: First submitted 2012-06-14; First posted 2012-06-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Tooth Erosion
Keywords: enamel erosion; ultrasound; reproducibility; human central incisor; reliability
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasound enamel thickness measurements (Other): Enamel thickness will be measured with ultrasound
  Interventions: Other: Ultrasound transducer

INTERVENTIONS:
Other: Ultrasound transducer — A hand-held ultrasound transducer will be placed on a central incisor and enamel thickness measurements recorded

SUMMARY:
The investigators have now established a technique to measure enamel thickness which has been shown to work well in-vitro. The teeth tested so far, obtained from the Dental School Tissue Bank, have been molars or pre-molars. In these cases, the measurement is made more difficult by the curvature of the tooth surface and it seems likely that flatter larger, incisors would give more satisfactory results. The investigators therefore wish to establish in-vivo whether this hypothesis is correct.

DETAILED DESCRIPTION:
The aim is translate our research into a clinical hand-held dental tool that could be used to measure enamel thickness in less curvaceous anterior incisor (front) teeth, and ultimately monitor erosive tooth surface loss (TSL), which mainly occurs on anterior (front) teeth and the occlusal (top) surface of posterior (back) teeth. In this study, quantifying enamel thickness with ultrasound will provide data which will be assessed for reproducibility and to determine whether or not ultrasound is a potentially viable tool to measure and monitor acid erosion of teeth. This would allow dentists to reinforce advice to patients to reduce acidic consumption, and will motivate them to keep whatever is remaining of their 'precious' enamel tissue, which if lost, will necessitate fillings to be made. These fillings will require future repairs and possible remakes, as they have median survival rates of five years.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults over 18 years (females and males) with normal salivary flow.
2. Volunteers with absence of dental caries and/or periodontal disease on the maxillary incisors (upper front teeth) to be used in the study.
3. Volunteers should have sound maxillary incisors with no obvious cracks in the crown.
4. Volunteers who willingly signed an informed consent.
5. Volunteers who are willing to follow the research schedule for the period of the study.

Exclusion Criteria:

1. Volunteers with abnormal enamel on maxillary incisors assessed by visual inspection.
2. Volunteers with replaced enamel on maxillary incisors (eg fillings, crowns, bridges).
3. Volunteers who appear to have hypoplastic teeth as part of a syndrome, e.g. osteogenesis imperfect.
4. Volunteers having orthodontic appliances on front teeth, or presence of fixed or removable dentures (replacing missing front teeth).
5. Volunteers who have a complex dental history such as periodontitis, dentine sensitivity or salivary dysfunction.
6. Volunteers who have any condition could be expected to interfere with the volunteer's safety during the study.
7. Volunteers who demonstrate an inability to comply with study procedures.
8. Signed informed consent not obtained by the volunteer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Enamel thickness reproducibility measurements | 2 weeks
  To know if ultrasound can reliably and reproducibly measure enamel thickness in-vivo

SECONDARY OUTCOMES:
Enamel thickness reproducibility measurements on separate occasions | 2 weeks (concurrent with primary outcome)
  To investigate whether ultrasound can be used to reproducibly measure enamel thickness on human incisor teeth in vivo on three separate occasions

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Sindi, BDS, Principal Investigator — University of Leeds (Leeds Dental Instiitute); Lynn Gutteridge, BDS, MDS, FDS RCS, MRD RCS, Study Chair — University of Leeds (Leeds Dental Institute); Nigel Bubb, Bsc, PhD, Study Director — University of Leeds (Leeds Dental Institute); Anthony Evans, BSc, MSc, PhD, CSci, Study Director — University of Leeds (Department of Medical Physics, Leeds Institute of Genetics, Health and Therapeutics)
Locations (1):
- University of Leeds, Leeds Dental Institute (DenTCRU), Leeds, West Yorkshire, United Kingdom